CLINICAL TRIAL: NCT03051295
Title: The Influence of Different Formats for Presenting Diagnostic Test Results and Treatment Efficacy on Dentists' Understanding and on Their Reported Clinical Management.
Brief Title: Dentists' Understanding of Diagnostic Test Results and Treatment Efficacy.
Acronym: RCDENT2017
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Rio de Janeiro State University (Other)
Responsible Party: Principal Investigator, Paulo Nadanovsky, Prof. Dr., Rio de Janeiro State University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: riskcommunicationdentist2017
Record Dates: First submitted 2017-02-06; First posted 2017-02-13 (Actual); Last update posted 2017-02-13 (Actual); Status verified 2017-02

CONDITIONS: Health Education
Keywords: Communication Barriers; Persuasive Communication; Risk
MeSH Terms: conditions — Health Education

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Diagnostic percentages. (Active Comparator): Dentist receives diagnostic test results presented in conditional probabilities.
  Interventions: Other: Dental health information form
- Diagnostic frequencies (Experimental): Dentist receives diagnostic test results presented in natural frequencies.
  Interventions: Other: Dental health information form
- Treatment percentages. (Active Comparator): Dentist receives treatment efficacy presented in percentages.
  Interventions: Other: Dental health information form
- Treatment frequencies. (Experimental): Dentist receives treatment efficacy presented in natural frequencies.
  Interventions: Other: Dental health information form

INTERVENTIONS:
Other: Dental health information form — The format in which dentists receive information about diagnostic test results and efficacy of treatment.

SUMMARY:
There is little evidence on how best to present diagnostic and treatment effect information to dentists and whether this makes any difference to their understanding of the information given and clinical management. The objective of this study is to assess the influence of different formats for presenting diagnostic test results and treatment efficacy on dentists' understanding and on their reported clinical management. The hypothesis is that presenting diagnostic test and treatment effectiveness results using natural frequencies influences the threshold for treatment and improves interpretation of tests results compared to conditional probabilities and percentage differences. A group of dentists recruited from postgraduate courses were randomized to two of four arms, being two arms of a hypothetical realistic diagnostic scenario (a) and two arms of a hypothetical realistic treatment scenario (b): a1) diagnostic test results presented in conditional probabilities; a2) diagnostic test results presented in natural frequencies; b1) treatment efficacy presented in percentages; b2) treatment efficacy presented in natural frequencies. The main outcome measures were the correct answer as to whether disease was actually present (post-test probability) and the correct answer as the number of patients that would benefit from the treatment (efficacy). Secondary outcome measures included the decision whether to treat or not treat the hypothetical patient.

ELIGIBILITY:
Inclusion Criteria:

* Graduated dentist undergoing a postgraduate course in a public university in Rio de Janeiro.

Exclusion Criteria:

* None.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 101 (Actual)
Dates: Start 2016-06-08 (Actual); Primary Completion 2016-12-13 (Actual); Study Completion 2016-12-13 (Actual)

PRIMARY OUTCOMES:
The probability that a patient will have a dental cavity as assessed by a dentist. | Up to 20 minutes
  The assessement by the dentist was based on a questionnarie containing a clinical hypothetical situation and the result of a bite-wing radiographic exam.
The number of patients that will benefit from systemic antibiotics adjunct to periodontal treatment as assessed by a dentist. | Up to 20 minutes
  The assessement by the dentist was based on a questionnarie containing a clinical hypothetical situation and the information about the usual efficacy of systemic antibiotics adjunct to periodontal treatment.

SECONDARY OUTCOMES:
The number of dentists that would recommend the use of systemic antibiotics adjunct to periodontal treatment in the clinical management of a patient with periodontal disease. | Up to 20 minutes
  The recommendation by the dentist was based on a questionnarie containing a clinical hypothetical situation and the information about the usual efficacy of systemic antibiotics adjunct to periodontal treatment.

IPD SHARING:
Plan to Share IPD: No